CLINICAL TRIAL: NCT05855889
Title: Observational Study of the Management of Infants With Congenital CMV
Acronym: cCMVnet
Status: Recruiting | Type: Observational
Sponsor: St George's, University of London (Other)
Collaborators: European Society for Paediatric Infectious Diseases (Other)
Responsible Party: Sponsor
Other Study IDs: 2021.0118
Record Dates: First submitted 2023-04-05; First posted 2023-05-12 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-05

CONDITIONS: Congenital Cmv
MeSH Terms: conditions — Cytomegalovirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is an observational, prospective/retrospective multicentre, cohort study of children diagnosed with cCMV. This study will contribute to a wider study also recruiting participants in Europe and other countries worldwide. No investigations or treatment will be carried out that are not part of routine clinical practice. Infants with cCMV are routinely followed up from an infectious diseases, audiology, ophthalmology and neurodevelopmental perspective until approximately 6 years of age, or longer if there are ongoing issues. Some children will be retrospectively diagnosed with cCMV in later childhood. Recruitment can be from any centre that manages these patients and has agreed to participate in the study.

DETAILED DESCRIPTION:
Cytomegalovirus (CMV) is the most frequent cause of congenital infection worldwide, occurring in 0.2-2% of live births. It is also the most frequent cause of non-genetic hearing loss, and an important cause of neurodevelopmental delay. Clinical diagnosis of maternal infection during pregnancy is unreliable in most patients and laboratory diagnosis can be challenging, especially in non-primary infections. Screening of congenital CMV infection (cCMV) in newborns is not recommended in most countries and only targeted screening is performed in some cases (children who fail hearing screening or with abnormalities compatible with cCMV in physical exams).

The main focus of the study is to identify patient and treatment characteristics that are associated with outcome. This will allow improved patient care in the future.

ELIGIBILITY:
Inclusion Criteria: Patients of either sex that have been diagnosed with cCMV infection:

* Through confirmed detection of CMV in urine or saliva, by CMV-DNA PCR (or viral culture / Shell-vial) and/or CMV detection in blood or CSF by PCR within the first 21 days of life.
* Children with cCMV retrospectively diagnosis by positive CMV-DNA PCR in dried blood spots (DBS), collected within 21 days of life.
* Diagnosed by positive CMV-DNA PCR in dried umbilical cord blood or donated/stored umbilical cord blood sample
* Children whose parents give their informed consent to participate in the study
* Age less than 11 years old

Exclusion Criteria:

* Refusal to sign written informed consent of parents/ legal guardian.

Max Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children will be identified at their routine healthcare attendance at the specialist clinics for children with congenital CMV at one of the participating centres. The person with parental responsibility will be approached to be informed about the registry and to request consent, either by the cCMVNET clinician or a delegated research nurse.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-03-09 (Actual); Primary Completion 2031-03-30 (Estimated); Study Completion 2038-03-30 (Estimated)

PRIMARY OUTCOMES:
Measuring cases of cCMV in the UK | 15 years
  To analyze the epidemiology of children born with cCMV
Clinical characteristics | 15 years
  To analyze the clinical characteristic of children born with cCMV (measure is number of participants with hearing loss, retinitis, neurological abnormalities, skin rashes, or hepatosplenomegaly)
To evaluate risk factors in children with cCMV for long term sequelae | 15 years
  To measure the number of cases with abnormal brain imaging (cranial USS or MRI), hearing loss, retinitis or anaemia, leucopenia, thrombocytopenia, renal function or liver abnormalities at diagnosis
Adverse events | 15 years
  To document adverse events of different treatment strategies
To evaluate the prognostic value of microbiological variables | 15 years
  To measure the urine CMV viral load in cases at diagnosis who develop hearing loss
To evaluate the prognostic value of image findings | 15 years
  To measure the number of cases who have abnormal brain imaging (cranial USS or MRI) at diagnosis and develop hearing loss
To evaluate associated outcomes with different treatment strategies | 15 years
  To measure the number of cases treated with valganciclovir and the number of treated cases who need a treatment break

CONTACTS AND LOCATIONS:
Overall Officials: Simon Drysdale, MD, Principal Investigator — St George's, University of London
Locations (1):
- St George's University of London, London, United Kingdom